CLINICAL TRIAL: NCT05592912
Title: Safety and Preliminary Efficacy of Two Dose Levels of HydroLenz as a Protectant for Vitrectomy-Induced Lens Opacities in Subjects Undergoing Vitrectomy
Brief Title: Safety and Efficacy of HydroLenz for Vitrectomy-Induced Lens Opacities
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding Limitations
Sponsor: PromiSight, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HL-001
Record Dates: First submitted 2022-10-18; First posted 2022-10-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Pars Plana Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low dose HydroLenz treatment (Experimental)
  Interventions: Drug: HydroLenz Injection
- High dose HydroLenz treatment (Experimental)
  Interventions: Drug: HydroLenz Injection
- Control, i.e., no HydroLenz treatment (Placebo Comparator)
  Interventions: Other: No HydroLenz Injection

INTERVENTIONS:
Drug: HydroLenz Injection — The HydroLenz injection will be administered at the conclusion of the vitrectomy procedure on the operative day
  Arms: High dose HydroLenz treatment; Low dose HydroLenz treatment
Other: No HydroLenz Injection — No HydroLenz injection will be administered at the conclusion of the vitrectomy procedure on the operative day.
  Arms: Control, i.e., no HydroLenz treatment

SUMMARY:
The primary objective of this study is to provide safety data for two different dosages of HydroLenz. Secondary objectives are to provide preliminary data to determine whether HydroLenz has the same effect in humans as it does in the porcine model; to confirm the reliability of methods for evaluating lens opacity; and, to acquire information that can be used to design the pivotal study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race.
2. 65 years of age or older.
3. Study eye is phakic and scheduled for pars plana vitrectomy (23, 25, or 27 gauge) for epiretinal membrane or vitreomacular traction surgery.
4. Willingness and ability to comply with schedule for follow-up visits.
5. Subject understands the study requirements and the treatment procedures and provides signed, written informed consent obtained in accordance with the institutional review board (or ethics committee) requirements for this first-in-man early feasibility study.

Exclusion Criteria:

1. Aphakic or pseudophakic lens status in either or both eyes.
2. History of previous cataract surgery in either eye.
3. Evidence of congenital cataract.
4. Study eye with corneal opacity of one of the following LOCS III grades or condition that would confound the LOCS III grading results:

   1. Inability to grade opacities in the study eye with LOCS III at the baseline exam;
   2. Inability to dilate pupil to at least 6.0 mm;
   3. LOCS III grade ≥ 2 for nuclear opalescence, cortical lens opacities, or posterior subcapsular lens opacities in the study eye at baseline.
5. Diabetic retinopathy or macular edema in the study eye.
6. Retinal vascular disease or retinopathy in the study eye.
7. History of previous intravitreal injections in the study eye.
8. History of previous subconjunctival injections in the study eye.
9. History of previous radiation in the study eye.
10. History of systemic, periocular, inhaled, or chronic topical corticosteroids.
11. Previous laser prophylaxis for retinal tear/hole/lattice degeneration in the study eye.
12. Previous pneumatic retinopexy or retinal detachment repair in the study eye.
13. Previous vitrectomy in the study eye.
14. Previous laser treatment anywhere in the study eye (trabecular meshwork, iris, retina, macula).
15. Use of silicone oil, air or gas tamponade during the vitrectomy in the study eye prior to injection of the HydroLenz.
16. Use of binocular indirect ophthalmoscopy laser during the procedure (endolaser is permitted).
17. History of any previous ocular surgery in the study eye.
18. Any ocular trauma resulting in lens opacity or subluxation of the lens in the study eye.
19. Iatrogenic lens trauma during surgery prior to injection of the HydroLenz.
20. Surgical plan for the vitrectomy includes planned glaucoma filtering or tube-shunt procedure or any procedure affecting the lens.
21. Female patients who are pregnant or lactating or plan to become pregnant during the course of the study.
22. A known sensitivity to study medications for which no alternative medication can be - prescribed.
23. Presence or history of any other condition or finding that, in the investigator's opinion, makes the patient unsuitable as a candidate for the HydroLenz treatment or study participation or may confound the outcome of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Changes in Lens Opacities | Baseline and 6 Months
  The Lens Opacity Classification System, Version III (LOCS III) and the rate of lens related (cataract) surgery will be used to evaluate the lens opacities.
Evaluation of Changes in Lens Opacities | Baseline and 12 Months
  The Lens Opacity Classification System, Version III (LOCS III) and the rate of lens related (cataract) surgery will be used to evaluate the lens opacities.
Changes in BSCVA | Baseline and 6 Months
  Number of eyes losing more than 2 lines of BSCVA
Changes in BSCVA | Baseline and 12 Months
  Number of eyes losing more than 2 lines of BSCVA

IPD SHARING:
Plan to Share IPD: No